CLINICAL TRIAL: NCT00270400
Title: Natrecor (Nesiritide) Versus Dobutamine Therapy for Symptomatic, Decompensated CHF: A Safety Study Using 24-Hour Holter Monitoring - The PRECEDENT Trial: Prospective, Randomized Evaluation of Cardiac Ectopy With Dobutamine or Natrecor Therapy
Brief Title: A Safety Study Comparing Natrecor (Nesiritide) Versus Dobutamine Therapy for Worsening Congestive Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scios, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005200
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Heart Failure, Congestive
Keywords: Heart Failure; Renal Dysfunction; Cardiomyopathy; Heart Decompensation; Dyspnea Paroxsymal.
MeSH Terms: conditions — Heart Failure; Renal Insufficiency; Cardiomyopathies | interventions — Natriuretic Peptide, Brain

ARMS (1):
- 001 (Experimental): nesiritide
  Interventions: Drug: nesiritide

INTERVENTIONS:
Drug: nesiritide

SUMMARY:
The purpose of this study is to compare the effects on heart rate and ventricular arrhythmias (irregular heart beats) of two doses of NatrecorÂ® (a recombinant form of the natural human peptide normally secreted by the heart in response to heart failure) versus dobutamine, during the first 24 hours of treatment of decompensated congestive heart failure (CHF).

DETAILED DESCRIPTION:
Advanced congestive heart failure (CHF) accounts for over one million hospital admissions yearly in the U.S. and is associated with a 2-year mortality rate of up to 40% - 50% (according to the American Heart Association 1997 and the CONSENSUS Trial Study Group, 1987). Inpatient therapy for acutely worsening CHF often includes intravenous (IV) agents to reduce intracardiac filling pressures and to increase cardiac output. Examples of such agents include drugs that increase the heart muscle contractility such as dobutamine and phosphodiesterase inhibitors such as milrinone. While these agents do achieve good blood flow throughout the body in most patients, several studies suggest that arrhythmias (irregular heart beats) can be increased in some patients treated with dobutamine or milrinone (according to Smith TW, et al 1997 and Holmes JR et al 1985; and Anderson JL et al 1986). Arrhythmias are common in patients with advanced CHF and may contribute to their sudden death rate of 30% to 70% (according to Stevenson WG, et al 1993).

Holter monitoring of patients with CHF shows 90% have premature ventricular contractions and non-sustained ventricular tachycardia (rapid beating) show up in 60% of patients (according to Stevenson WG, et al 1994) and atrial fibrillation in approximately 20% of patients (according to Smith TW, et al 1997). The occurrence of arrhythmias may be associated with a decrease in ventricular performance, which may worsen the symptoms of acutely decompensated CHF and complicate patient management. The ventricle is the heart's pumping chamber that pumps the oxygen-poor blood returning from the body into the arteries of the lungs, where the blood picks up oxygen. In atrial fibrillation the heart's two small upper chambers (the atria) quiver instead of beating effectively. Therefore, it is imperative that new therapies developed for the treatment of decompensated CHF not be associated with the development or an increase of arrhythmias. Natrecor® has been studied as an IV treatment for decompensated CHF in over 500 patients. As interstitial fluid (in the lung tissues) accumulates in advanced CHF cases, the pulmonary capillary wedge pressure (PCWP) increases. However administration of a continuous IV infusion of Natrecor® resulted in dose-related decreases in PCWP, right atrial pressure, and systemic vascular resistance, and an increase in cardiac index which is a measurement of the volume of blood pumped by the heart, (according to Marcus LS, Hart D, Packer M, et al 1996; Abraham WT at al 1998; and Mills RM et al 1999 ). Beneficial improved blood flow throughout the body associated with a decrease in the systolic blood pressure - heart rate index (the double product), suggests that Natrecor® improves cardiac performance while not increasing estimated myocardial oxygen consumption.

The primary objective of this study is to compare the effects on heart rate and ventricular arrhythmias of two doses of Natrecor® to dobutamine, during the first 24 hours of treatment of decompensated CHF. The primary outcome of the study is an evaluation of: (1) average heart rate, (2) average hourly premature ventricular beats, and (3) average hourly repetitive beats, all expressed as a change from baseline, as measured by Holter monitoring (a portable device that provides continuous monitoring of the electrical activity of the heart). Additional objectives include exploring the effects of Natrecor® and dobutamine on other Holter outcomes such as couplets, triplets, and ventricular tachycardia and the evaluation of ventricular ectopy (seven or more single premature ventricular beats per minute or any run of more than two ventricular ectopic beats) by the application of specific proarrhythmic criteria. Clinical symptoms are also measured.

This is a multicenter, randomized, open-label, active-controlled safety study designed to enroll approximately 240 patients with symptomatic (New York Heart Association [NYHA] Class III or IV), decompensated CHF for whom treatment with dobutamine or Natrecor® is deemed appropriate. After a 24-Hour Baseline Holter Monitoring Period, patients are randomized to dobutamine or Natrecor® (0.015 or 0.03 µg/kg/min). The randomization is stratified by whether or not the subjects have a known history of Ventricular Tachycardia (non-sustained or sustained). Treatment assignment is open-label with regard to the study drug (dobutamine or Natrecor®); assignment to the two Natrecor® dose groups is double-blinded. Dobutamine is to be administered at a dose of at least 6 µg/kg/min. During the first 24 hours of study drug, each patient undergoes Holter monitoring. Study drug (dobutamine or Natrecor®) is administered for at least 24 hours as the single IV vasoactive agent for symptomatic, decompensated CHF. Other IV vasoactive agents such as milrinone, nitroprusside, nitroglycerin, and/or any dose of dopamine are not to be added to the study drug during the first 24 hours of therapy. Dobutamine is not to be added to the Natrecor® infusion during the first 24 hours of therapy. After 24 hours, the Holter monitor will be removed, and patients can remain on study drug, if appropriate. Natrecor® patients can continue on their fixed-dose Natrecor® regimens (still blinded to specific dose group assignment) for up to a maximum of 7 days (with or without the addition of other parenteral agents) or can switch to whatever treatment is appropriate, at the discretion of the investigator. Patients in the dobutamine treatment group can continue on study drug as long as appropriate, at the discretion of the investigator. Systemic hemodynamics (blood pressure and heart rate) are assessed at baseline, at 15 and 30 minutes, and at 3, 8, 16, and 24 hours following the initiation of study drug. The study hypothesis is that Natrecor® is not associated with increases in reported ventricular arrhythmias in patients being treated for symptomatic decompensated CHF. Continuous IV (intravenous) Infusion for at least 24 hours, and over 24 hours with discretion of Principal Investigator. Dobutamine starts at 5 mcg/kg/min, may be increased; Natrecor®, either 0.015 mcg/kg/min or 0.030 mcg/kg/min fixed dose for at least 24 hours, up to a maximum of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* History of NYHA (New York Heart Association) Class III or IV congestive heart failure (CHF)
* Has symptomatic, decompensated CHF for which inpatient therapy with either dobutamine or Natrecor®, administered as a single intravenous vasoactive agent (drugs that influence the tone and caliber of blood vessels) with or without diuretics, is deemed appropriate
* Receiving stable doses of oral antiarrhythmic medications (medications that help regulate irregular heart beats) for at least the 48 hours before starting study drug, or receiving no antiarrhythmic medications.

Exclusion Criteria:

* Cannot tolerate a 24-Hour Baseline Holter Monitoring Period without intravenous vasoactive medications, and/or cannot tolerate the specified washout period (if applicable) of intravenous vasoactive medications before starting the baseline Holter monitoring
* Has systolic blood pressure consistently < 85 mm Hg, cardiogenic shock, or other evidence of significant hemodynamic instability requiring the immediate institution of inotropic/pressor support
* Has a clinical condition expected to require therapy with more than one intravenous vasoactive agent or Dopamine during the 24-Hour Treatment Holter Monitoring Period
* Has received treatment with Dopamine or any intravenous vasoactive medication such as Dobutamine, Milrinone, Nitroprusside or intravenous Nitroglycerin for more than 4 hours for the current episode of decompensated CHF or related illness
* Requires an intravenous antiarrhythmic medication during the 48 hours before starting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 1998-08; Study Completion 1999-02 (Actual)

PRIMARY OUTCOMES:
Average heart rate; average hourly premature ventricular beats; average hourly repetitive beats, all expressed as a change from baseline

SECONDARY OUTCOMES:
Incidence of tachycardia through 24 hours; Incidence of tachycardia, pain, and injection site reaction through 14 days .

CONTACTS AND LOCATIONS:
Overall Officials: Scios, Inc. Clinical Trial, Study Director — Scios, Inc.

REFERENCES:
- [Result] Burger AJ, Horton DP, LeJemtel T, Ghali JK, Torre G, Dennish G, Koren M, Dinerman J, Silver M, Cheng ML, Elkayam U; Prospective Randomized Evaluation of Cardiac Ectopy with Dobutamine or Natrecor Therapy. Effect of nesiritide (B-type natriuretic peptide) and dobutamine on ventricular arrhythmias in the treatment of patients with acutely decompensated congestive heart failure: the PRECEDENT study. Am Heart J. 2002 Dec;144(6):1102-8. doi: 10.1067/mhj.2002.125620. PMID 12486437
- [Derived] Nearing BD, Wellenius GA, Mittleman MA, Josephson ME, Burger AJ, Verrier RL. Crescendo in depolarization and repolarization heterogeneity heralds development of ventricular tachycardia in hospitalized patients with decompensated heart failure. Circ Arrhythm Electrophysiol. 2012 Feb;5(1):84-90. doi: 10.1161/CIRCEP.111.965434. Epub 2011 Dec 8. PMID 22157521